CLINICAL TRIAL: NCT04999319
Title: Comparison of Morphine Consumption at Postoperative 24th Hour in Thoracotomy: A Randomized Controlled Trial
Brief Title: Morphine Consumption in Thoracotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Mustafa Duran, MD, Principal investigator., Kocaeli University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: GOKAEK-2020/18.09
Record Dates: First submitted 2021-08-05; First posted 2021-08-10 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Postoperative Pain
Keywords: Postoperative pain; Thoracotomy; Paravertebral block; Erector spina plane block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PVB Group (Active Comparator): Paravertebral block administered group
  Interventions: Procedure: PVB
- ESPB group (Active Comparator): Erector spinae plane block administered group
  Interventions: Procedure: ESPB

INTERVENTIONS:
Procedure: PVB — Paravertebral block will be performed before the surgery with 20 mL of %0.5 bupivacaine at T4 level.
  Arms: PVB Group
Procedure: ESPB — Erector spinae plane block will be performed before the surgery with 20 mL of %0.5 bupivacaine at T4 level.
  Arms: ESPB group

SUMMARY:
Importance of effective postoperative pain management is well known. The undesired effects of pain can be prevented with multimodal analgesia for the patient. Thoracotomy operations are associated with high levels of pain. With the use of ultrasound, many regional anesthesia techniques were described to provide effective postoperative analgesia. The aim of this study was to compare the postoperative effect of paravertebral block (PVB) and erector spinal plane block (ESPB) in thoracotomies.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III patients undergo elective thoracotomy surgeries.

Exclusion Criteria:

* Obesity (BMI > 35 kg/m2)
* Infection of the skin at the site of the needle puncture area
* Patients with known allergies to any of the study drugs
* Coagulopathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | Postoperative 24th hour
  Morphine consumption (mg) of patients with patient controlled analgesia device
NRS score | Postoperative 24th hour
  Numerating rating scale of the patients (between 0 and 10, 0 represents no pain and 10 represents the worst pain ever possible.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli Unversity, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No